CLINICAL TRIAL: NCT03983018
Title: Rituximab - Immunotherapy for Schizophrenia Spectrum Disorder in Adults: An Open Pilot Study
Brief Title: Rituximab for Schizophrenia Spectrum Disorder (RITS-PS-2019)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Susanne Bejerot, Professor, Region Örebro County
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Number: 2018-004618-17
Record Dates: First submitted 2019-05-30; First posted 2019-06-12 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders; Treatment-resistant Schizophrenia
Keywords: Immunopsychiatry; Schizophrenia spectrum disorder; treatment-resistant
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Schizophrenia, Treatment-Resistant | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: open trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental): 1000 mg of rituximab, infusion once
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Infusion

SUMMARY:
This study evaluates the addition of rituximab to 12 patients diagnosed with treatment resistant schizophrenia spectrum disorder in an open trial.

DETAILED DESCRIPTION:
Immunological factors may be determinants for some psychiatric disorders, thus immunomodulation may be helpful. Rituximab (antibodies against CD20, cluster of differentiation), a standard treatment for multiple sclerosis, is an anti-inflammatory drug, hitherto not tested for psychiatric disorders.

The aim of this study is to investigate whether the psychiatric symptoms of treatment-resistant adult psychiatric patients, diagnosed with schizophrenia spectrum disorder (SSD), are significantly improved after treatment with rituximab. Our purpose is to implement recent insights from "Immunopsychiatry" to find efficacious, but still tolerable treatment for these patients.

This is a single-site, 20-week, open pilot, add-on treatment as usual, trial, where the patients will be followed for 1 year.

Rituximab will be administered with one single dose of 1000 mg. Investigators will analyse inflammatory and metabolic biomarkers in relation to the primary outcome, treatment response (defined as clinically relevant reduction in the validated measure PANSS). Other outcomes are "much" or "very much improved" on Clinical Global Impression - Improvement scale (CGI-I) and change in Personal and Social Performance Scale measuring overall disability.

ELIGIBILITY:
Inclusion Criteria (Swedish citizens):

1. patient ages 18 to 40 years
2. a duration of illness exceeding 2 years
3. correspond to "Markedly ill", "Severely ill" or "Among the most extremely ill patients" on the Clinical Global Impression - Severity scale (CGI-S)
4. Global Assessment of Functioning below 50
5. Schizophrenia spectrum disorder according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
6. treatment resistance, i.e. failing to remit despite adequate treatments
7. if female and with any risk for pregnancy, willing to use contraceptives
8. if antipsychotic treatment is prescribed the plasma concentrations of the drug must be tested and shown to be within therapeutic interval.
9. subjects should be judged by the investigator to be lucid and oriented to person, place, time, and situation when giving the informed consent.
10. immunoglobulin levels within the normal range

Exclusion Criteria:

1. on-going immunomodulatory treatment
2. pregnancy or breast-feeding
3. weight below 40 kg
4. clinically relevant on-going infection
5. chronic infections
6. positive screening test for hepatitis B, C, HIV or tuberculosis
7. any change of psychotropic medication within the previous 4 weeks
8. "much" or "very much improved" already at baseline according to CGI-I i.e. scores of 1 or 2 by the clinician
9. severe heart failure (NYHA grade IV) or other severe heart disease or history of cardiac arrhythmia or myocardial infarction
10. unable to make an informed decision to consent to the trial
11. in compulsory treatment
12. treatment with clozapine within the last 2 months
13. previous treatments with immunosuppressive agents
14. malignancy currently or within 2 years prior to inclusion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bejerot, Principal Investigator — Region Orebro lan
Locations (1):
- Region Örebro Län, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No
Details that can identify the patients will not be shared.

REFERENCES:
- [Result] Bejerot S, Sigra Stein S, Welin E, Eklund D, Hylen U, Humble MB. Rituximab as an adjunctive treatment for schizophrenia spectrum disorder or obsessive-compulsive disorder: Two open-label pilot studies on treatment-resistant patients. J Psychiatr Res. 2023 Feb;158:319-329. doi: 10.1016/j.jpsychires.2022.12.003. Epub 2022 Dec 20. PMID 36638622
- [Result] Thunberg P, Fresnais D, Hamilton P, Bejerot S, Humble MB. Immunomodulatory treatment may change functional and structural brain imaging in severe mental disorders. Brain Behav Immun Health. 2024 Sep 16;41:100864. doi: 10.1016/j.bbih.2024.100864. eCollection 2024 Nov. PMID 39350952

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Pilot: 9 patients reached 12 weeks of treatment. 8 reached endpoint I at 20 weeks and endpoint II 40 weeks.
Period: Overall Study
Arm/Group | Open Pilot
Started | 9
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Rituximab: 1000 mg rituximab infusion once
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — white
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 9
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Local psychiatrists were invited to include patients and we also recruited through patient organisations
  participants
    Sweden | 9
Positive and Negative Syndrome Scale (PANSS) [Mean (Standard Deviation); unit: units on a scale] — standarised interview with Positive and Negative Syndrome Scale (PANSS)
  units on a scale | 99 (32)
The Personal and Social Performance Scale (PSP) [Mean (Standard Deviation); unit: units on a scale] | 32.0 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: Change in symptoms measured as change in Positive and Negative Syndrome Scale (PANSS) score from baseline. PANSS measures symptom severity of patients with schizophrenia and is a clinically based interview. PANSS measures positive symptoms (7 items, range 7-49), which refer to e.g. hallucinations and delusions; negative symptoms (e.g. loss of normal functions) (7 items, range 1-7) and general disability (16 Items, range 16 -112) separately. Higher scores denote more symptoms and disability. PANSS total score range from 30-210. At least 40 % reduction in PANSS total score is regarded as response.
Time Frame: week 20
Population: Eight patients reached week 20.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Rituximab 1000 mg infusion once
Arm/Group | Experimental
Number analyzed (Participants) | 8
score on a scale | 72.9 (36.2)

2. Secondary Outcome: Personal and Social Performance Scale (PSP)
Description: Personal and Social Performance Scale (PSP) gives a score for disability. The PSP is a 100-point single-item rating scale (range 1-100), subdivided into 10 equal intervals. Lower scores denote lower functioning. The ratings are based mainly on the assessment of patient's functioning in four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours. Change in score between enrolment and week 20 will be measured.
Time Frame: week 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental
Number analyzed (Participants) | 8
score on a scale | 53.1 (22.2)

3. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Scale
Description: CGI-S is a clinician rated measure of overall clinical severity that is rated on a scale between 1 and 7. A person with no clinical complaints or problems will get a score of 1. The score 7 indicates the highest level of severity is phrased as "Among the most extremely ill patients".
Time Frame: week 20
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) in Relation to Inflammatory Markers
Description: Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Change in inflammatory markers in blood (gene expression and proteins) towards normality, in relation to clinical response will be measured.
Time Frame: week 20
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I). Proportion of Responders.
Description: Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. If the mean value of these three is below 2.5 then the patient will be regarded as a responder (representing much or very much improved since baseline).
Time Frame: week 20
Reporting Status: Not Posted

6. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I).
Description: Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. Range 3-21. A lower score depicts larger improvement.
Time Frame: week 20
Reporting Status: Not Posted

7. Secondary Outcome: Adverse Event: Any Adverse Reactions (AAR). Safety and Tolerability of Rituximab
Description: Any Adverse reactions (AAR) is a rating scale developed for this study and is not a validated questionnaire. It consists of a list of 26 symptoms. AAR maps adverse events related to rituximab treatment. These items are assessed for severity on a Likert scale (4 levels: none; mild; moderate; severe) and frequency (3 levels: occasionally; daily; several times daily). AAR is assessed by the clinician. An adverse event scale was required as an outcome measure by the Swedish Medical Products Agency.
Time Frame: week 20
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: as for outcome 1
Time Frame: week 40
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Personal and Social Performance Scale (PSP)
Description: Personal and Social Performance Scale (PSP) gives a score for disability. The PSP is a 100-point single-item rating scale (range 1-100), subdivided into 10 equal intervals. Lower scores denote lower functioning. The ratings are based mainly on the assessment of patient's functioning in four main areas: 1) socially useful activities; 2) personal and social relationships; 3) self-care; and 4) disturbing and aggressive behaviours. Change in score between enrolment and week 40 will be measured.
Time Frame: week 40
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Clinical Global Impression-Severity (CGI-S) Scale
Description: Clinical Global Impression-Severity (CGI-S) scale is a clinician rated measure of overall clinical severity that is rated on a scale between 1 and 7. A person with no clinical complaints or problems will get a score of 1. The score 7 indicates the highest level of severity is phrased as "Among the most extremely ill patients".
Time Frame: week 40
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Clinical Global Impression-Improvement (CGI-I) in Relation to Inflammatory Markers
Description: Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Change in inflammatory markers in blood (gene expression and proteins) towards normality, in relationship to clinical response Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Change in inflammatory markers in blood (gene expression and proteins) towards normality, in relation to clinical response (assessed by the clinician) will be measured.
Time Frame: week 40
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in Cognitive Functioning
Description: The clinical assessment includes four sections of the Wechsler intelligence scales for adults (WAIS-IV); block design (range 1-19), letter number sequencing (range 1-19), digit symbol coding (range 1-19), and digit span (range 1-19). A full scale IQ of each participant will be estimated using the mean of the four scaled scores available and multiplying them by 11. A higher score denotes a cognitive improvement.
Time Frame: week 20
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Clinical Global Impression-Improvement (CGI-I).
Description: Clinical Global Impression-Improvement scale (CGI-I) measures change of symptoms on a 7 point Likert scale. A CGI-I score of 1 or 2 corresponds to be much or very much improved. Three different informants base their CGI-I evaluations on independent assessments: a) The treating clinician, b) The patient's self-assessment and c) A next of kin. If the mean value of these three is below 2.5 then the patient will be regarded as a responder (representing much or very much improved since baseline). Range 3-21. A lower score depicts larger improvement.
Time Frame: week 40
Reporting Status: Not Posted

14. Other Pre Specified Outcome: B-cell Subpopulations in Relation to Clinical Response
Description: B-cell depletion at week 5, and B-cell subpopulations at week 20 in relation to clinical response (CGI-I) (assessed by the clinician) and baseline levels of B-cells.
Time Frame: week 20
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Life Quality Measured With Brunnsviken Brief Quality of Life Scale (BBQ)
Description: BBQ is a 12-item self-rated measurement of life satisfaction. BBQ is a Likert scale, range 0-48. Higher scores denote higher life satisfaction.
Time Frame: week 40
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Clinical Global Impression-Improvement (CGI-I). Proportion of Responders.
Description: as for outcome 5
Time Frame: week 40
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Rituximab: Rituximab 1000 mg infusion once
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=9)
Abdominal Pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=9)
Long term covid (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03983018/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03983018/ICF_001.pdf